CLINICAL TRIAL: NCT03464240
Title: Investigating the Molecular Mechanisms Underpinning Glucose Stimulated Release of Stored Enteral Lipid in Humans
Brief Title: Glucose-stimulated Gut Lipid Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Kensington Screening Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Glucose Biopsy 15-9025
Record Dates: First submitted 2018-02-09; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — Glucose; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose (Active Comparator): 50 grams glucose in 50 ml water
  Interventions: Dietary Supplement: Glucose
- Water (Placebo Comparator): 50 ml water
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Glucose — glucose drink
  Arms: Glucose
Dietary Supplement: Water — control
  Arms: Water

SUMMARY:
During dietary fat absorption, the gut packages the majority of the fats into lipid particles that are secreted into blood circulation. The gut is also capable of storing a considerable amount of fats that can be released at a later time upon receiving certain stimulus signals. One of the signals is glucose ingestion. This protocol examines how glucose ingestion releases gut lipid store. Participants drink a fatty formula and 5-9 hours later drink either a glucose solution or water (as control). One hour later, duodenal biopsy specimen are taken for analysis of lipid stores in the gut cells.

DETAILED DESCRIPTION:
Participants undergoing upper gastrointestinal endoscopy and duodenal biopsy for clinical indications are recruited after obtaining informed consent. They first have a high fat liquid formula. 5 to 9 hours later, half of the participants drink 50 grams of glucose in 50 ml of water. The other half drink 50 ml of water. 1 hour later, duodenal biopsy specimen are collected and stored for analysis of lipid stores in the gut using electron microscopy and proteins using proteomics.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 60 years requiring endoscopy and duodenal biopsies for clinical indications, with no contraindications to the procedure, as judged by endoscopy doctor.
* Body mass index 20 to 27 kg/m2

Exclusion Criteria:

* Patients with active inflammatory bowel disease
* Patients with Celiac disease, exocrine pancreatic insufficiency or small bowel malabsorption
* Patients with active bowel malignancy
* Patients with diabetes mellitus or known/ suspected motility disorders of the gut
* Patients with decompensated liver disease
* Patients on ezetimibe or bile acid sequestrants
* Unstable cardiac or respiratory disease
* Any changes to medication in the preceding month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Visualization of lipid stores in the gut | 6-10 hours
  Electron microscopy observation gut samples in response to glucose versus water drink

SECONDARY OUTCOMES:
Analysis of proteins in the gut | 6-10 hours
  Proteomics analysis of gut samples in response to glucose versus water drink

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Tornto General Hospital, UHN, Toronto, Ontario
  - Kensington Screening Clinic, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No